CLINICAL TRIAL: NCT03462459
Title: Efficacy of Oral Vancomycin Prophylaxis for Prevention of Recurrent Clostridium Difficile Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical College of Wisconsin (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Henry Ford Hospital (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-0927; 1R01HS025713-01 (AHRQ); A534265 (Other: UW, Madison); SMPH/MEDICINE/INFECT DIS (Other: UW, Madison); Protocol ver 6, 18 Nov 2020 (Other: UW Madison)
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Clostridium Difficile Infection; Clostridium Difficile Infection; CDI; C.Difficile Diarrhea; C. Diff Colitis; C.Difficile Colitis
Keywords: Oral vancomycin; vancomycin; antibiotic
MeSH Terms: conditions — Clostridium Infections; Enterocolitis, Pseudomembranous | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin (Experimental): 125 mg, oral capsule by mouth, once daily, for the duration of standard-of-care antibiotic therapy plus 5 days
  Interventions: Drug: Vancomycin
- Placebo (Placebo Comparator): 125 mg placebo capsule by mouth, once daily, for the duration of standard-of-care antibiotic therapy plus 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vancomycin — Vancomycin capsule, 125 mg
  Other Names: Vancomycin Hydrochloride; Vancocin
  Arms: Vancomycin
Drug: Placebo — Capsule containing inert (nonactive) material to mimic 125 mg vancomycin capsule
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of prophylaxis with oral vancomycin for preventing recurrent Clostridium difficile Infection (CDI) in patients who have experienced at least one CDI episode in the last 180 days and are receiving antibiotics for a non CDI condition. Participants will be randomized to receive either placebo or oral vancomycin in addition to their prescribed antibiotic therapy.

DETAILED DESCRIPTION:
Many patients who have a CDI experience recurrent or relapsing symptoms. The investigators are studying whether vancomycin in low doses will help prevent further CDI episodes and how this therapy impacts patients' gastrointestinal microbiome and composition.

Patients with a history of past CDI who are receiving antibiotics for a non-CDI condition will be invited to participate. Approximately half of the participants will receive a low-dose capsule of vancomycin and half will receive a placebo. Participants will continue taking the vancomycin/placebo for 5 days after their prescribed antibiotics end.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent.
* Willing to comply with all study procedures and be available for the duration of the study.
* Documented diagnosis of at least one CDI within the last 180 days with treatment completed.
* Currently receiving systemic antibiotics for a non-CDI condition with anticipated duration of no more than 2 weeks.
* Females of childbearing potential must have a negative pregnancy test prior to randomization and agree to use adequate contraception prior to randomization, for the duration of the study, and for 4 weeks following study completion.
* Have received no more than 72 hours of non-CDI antibiotics.

Exclusion Criteria:

* History of hypersensitivity or allergy to oral vancomycin.
* Current use of oral vancomycin
* Patients on concurrent treatment with metronidazole or tetracycline monotherapy for any indication
* Patients diagnosed with inflammatory bowel disorder (Crohn's disease), or bacterial gastrointestinal infection cause by agents other than C. difficile (e.g. Salmonella sp.), toxic megacolon and/or known small bowel ileus.
* Dysphagia (inability to swallow capsules) or unwilling to swallow capsules.
* Major gastrointestinal surgery within 3 months of enrollment (does not include appendectomy or cholecystectomy).
* Any history of total colectomy or bariatric surgery.
* Unable or unwilling to fulfill study requirements.
* Expected life expectancy < 6 months.
* Patients enrolled in another clinical trial with investigational drugs within 30 days prior to randomization.
* Women who are pregnant or breast-feeding.
* Any patient deemed not suitable for study participation at the discretion of the study investigator.
* Diarrhea (3 or more loose stools in a 24 hour period) at enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Keating JA, Xu T, Graham MB, Ramesh M, Khanna S, Dixon J, Kates A, Haight K, Zhao J, Saddler C, Safdar N. Oral Vancomycin for Prevention of Recurrent Clostridioides difficile Infection: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2517834. doi: 10.1001/jamanetworkopen.2025.17834. PMID 40601321

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vancomycin | Placebo
Started | 37 | 42
Completed | 30 | 29
Not Completed | 7 | 13
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Unable to complete doses of study drug/placebo | 0 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Unable to obtain stool samples at visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: Adults age 18 or older with a diagnosis of recurrent Clostridioides diffcile infection
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin | Placebo | Total
Number analyzed (Participants) | 37 | 42 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.89 (15) | 58.40 (13) | 58.65 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 13 | 17 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 36 | 40 | 76
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 42 | 79

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Clostridium Difficile Infection (CDI)
Description: Determine whether CDI recurrence is decreased in patients taking oral vancomycin as prophylactic therapy in addition to standard-of-care antibiotics that patients are taking for non-CDI reasons.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 37 | 42
Participants | 17 | 24
Statistical Analysis 1: Comparison: Vancomycin vs Placebo; Test type: Equivalence — Proportional tests (Chi-squared) compared the episodes of C. difficile. Log-rank tests (Kaplan-Meier) were conducted to compare the non-recurrence proportions within the eight-week period. Multivariate Cox proportional hazard regression determined if treatment, age, and number of previous C. difficile episodes were predictors of recurrence; p = 0.22, Chi-squared; See comments = -0.11, 95% CI 2-sided [-35.1 to 8.0] — Proportional tests compared episodes of C. difficile recurrence in eight weeks (vancomycin vs. placebo) using Chi-squared test. Log-rank tests compared the non-recurrence proportions within 8 weeks with the Kaplan-Meier method; Statistical analyses are primarily reported for the population who were randomized in the study ("as randomized"). The secondary statistical analyses are reported for the population who completed all three visits ("as completed treatment"). Proportional tests were conducted to compare the episodes of C. difficile recurrence in eight weeks following the completion of the study intervention in patients receiving vancomycin versus placebo using the Chi-squared test. Log-rank tests were conducted to compare the non-recurrence proportions within the eight-week period in patients receiving vancomycin versus placebo with the Kaplan-Meier method. A nonparametric Wilcoxon rank sum test was used to compare distributions of the number of days to the first recurrence of CDI after starting oral vancomycin or placebo. The significance level was set to be ≤0.05. All statistical analyses were conducted in R statistical software (version 4.4.0; R Core Team, 2024)

2. Secondary Outcome: Gut Microbiome Composition
Description: Study how the gut microbiome is altered in patients receiving vancomycin treatment compared to placebo.
Time Frame: 8 weeks
Measure: Count of Units; unit: stool samples
Units Other Than Participants: stool samples
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 39 | 42
Number analyzed (stool samples) | 39 | 42
stool samples | NA — Data could not be reported due to low sample volumes for genomic sequencing. Genomic sequencing could not be done and comparisons between vancomycin and placebo also cannot be done. | NA — Data could not be reported due to low sample volumes for genomic sequencing. Genomic sequencing could not be done and comparisons between vancomycin and placebo also cannot be done.

3. Secondary Outcome: Vancomycin-resistant Enterococcus (VRE) Colonization in Stool Samples of Patients Receiving Vancomycin vs. Patients Receiving Placebo
Description: Low-dose exposure to vancomycin and VRE infection has not been studied. We will examine the incidence of VRE colonization in stool samples of all patients and determine whether oral vancomycin increases the VRE colonization rate, which has a negative impact on the overall health of patients being treated with vancomycin for C. difficile infection.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 37 | 42
Participants | 15 | 6
Statistical Analysis 1: Comparison: Vancomycin vs Placebo; Test type: Equivalence — Proportional difference tests comparing the proportion of patients with VRE colonization at Visit 3, compared to baseline. Significance level was set to 0.10; p = 0.10, Proportional difference test

4. Secondary Outcome: Determine Whether Clostridium Difficile Positivity on Any Stool Sample is a Predictor of CDI Recurrence.
Description: Stool samples will be tested at baseline, at the last dose date of vancomycin or placebo, at approximately 8 weeks following the last dose of vancomycin or placebo, and as indicated for diarrhea symptoms. Samples will be collected and tested for the presence of Clostridium difficile.
Time Frame: 8 weeks
Measure: Count of Units; unit: stool samples
Units Other Than Participants: stool samples
Arm/Group | Vancomycin | Placebo
Number analyzed (Participants) | 39 | 42
Number analyzed (stool samples) | 39 | 42
stool samples | NA — Data cannot be reported due to low available sample volumes for culture testing. | NA — Data cannot be reported due to low available sample volumes for culture testing.

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Vancomycin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/37 | 2/42
Serious Adverse Events (participants affected / at risk) | 9/37 | 10/42
Other Adverse Events (participants affected / at risk) | 37/37 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin (N=37) | Placebo (N=42)
Pneumonia with associated shock (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia/Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Elevated liver function tests due to transplant (Gastrointestinal disorders) | 1 (3) | 0 — Elevated liver function tests secondary to transplant
Recurrent C difficile Infection (rCDI) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0
Sickle Cell Pain Crisis (Blood and lymphatic system disorders) | 1 (4) | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) — Right arm
Thrombophlebitis (Infections and infestations) | 0 | 1 (1) — Right arm
Nausea (Gastrointestinal disorders) | 0 | 1 (1) — Post chemotherapy
Vomiting (Gastrointestinal disorders) | 0 | 1 (1) — Post chemotherapy
Nausea (Gastrointestinal disorders) | 0 | 1 (1)
Congestive Heart Failure Exacerbation (Cardiac disorders) | 1 (1) | 0
Whipple Procedure (Surgical and medical procedures) | 1 (1) | 0 — Planned hospitalization for procedure
General weakness/malaise (General disorders) | 0 | 1 (1) — Hospitalization due to general weakness/malaise
Toe Infection (Infections and infestations) | 1 (1) | 0
Osteomyelitis (Infections and infestations) | 1 (1) | 0
Altered Mental Status (Psychiatric disorders) | 0 | 1 (1) — Multifactorial Altered Mental Status
Traumatic fall with sequelae (Injury, poisoning and procedural complications) | 0 | 1 (1)
Carotid endarctectomy with stents (Vascular disorders) | 0 | 1 (1)
Peripheral autologous stem cell transplant (Surgical and medical procedures) | 0 | 1 (1) — Planned procedure due to stem cell transplant
Sigmoid resection surgery (Surgical and medical procedures) | 0 | 1 (1) — Sigmoid resection due to diverticulitis
Vaginal Polyp (Reproductive system and breast disorders) | 0 | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1) | 0 — New onset ACC/AHA Stage C HFpEF
Urinary Tract Infection (Infections and infestations) | 0 | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1 (1) — Small bowel obstruction secondary to colon cancer
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vancomycin (N=37) | Placebo (N=42)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (8) | 10 (12) — Diarrhea
Fever/Flu-Like Symptoms (General disorders) | 3 (3) | 2 (2) — Fever/Flu-Like Symptoms
UTI (Infections and infestations) | 3 (4) | 1 (1) — Urinary tract infection
Infections (Infections and infestations) | 4 (5) | 3 (3) — Infections
Joint pain and swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) — Joint pain and swelling
Abdominal Pain/Discomfort (Gastrointestinal disorders) | 9 (12) | 9 (9)
Nausea/Vomiting (Gastrointestinal disorders) | 9 (10) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (6) | 8 (9)
Bloating/flatulence (Gastrointestinal disorders) | 4 (4) | 7 (7)
Bloody stool/loose stool (Gastrointestinal disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT03462459/Prot_SAP_007.pdf
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT03462459/ICF_008.pdf